CLINICAL TRIAL: NCT02175810
Title: Impact of Bariatric Surgery on Cardiorespiratory Function: an Observational Study
Brief Title: Impact of Bariatric Surgery on Cardiorespiratory Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St George's, University of London (Other)
Collaborators: Universidade Federal do Triangulo Mineiro (Other); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Sponsor
Other Study IDs: 13.0217
Record Dates: First submitted 2014-06-25; First posted 2014-06-26 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Obesity; Bariatric Surgery Candidate; Physical Activity
Keywords: Obesity; Bariatric surgery; physical activity; cardiopulmonary exercise test
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Obesity is a growing problem worldwide and its prevention has become one of the leading priorities for the World Health Organisation. Obesity results from chronic imbalance between energy intake and energy expenditure. Although early prevention of obesity is preferable, surgical treatment is often required for severely obese people.

Bariatric surgery has been shown to be the most effective therapy for severe obesity. Weight loss following bariatric surgery results in significant improvements in coexisting comorbidities, such as diabetes and hypertension but there is controversy whether bariatric surgery also improves aerobic capacity.

The purpose of this study is to investigate the effects of bariatric surgery on cardiopulmonary function and on daily physical activity. It is hypothesized that bariatric surgery will improve aerobic capacity and result in beneficial lifestyle changes from sedentary to more active.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 years to 50 years
* Patients enrolled in the bariatric surgery program of St George's Hospital with BMI > 40 kg/m2, or 35-40 kg/m2 in the presence of other obesity-related comorbidities such as hypertension or type- 2 diabetes

Exclusion Criteria:

* Locomotor difficulties which would prevent participants from completing the cardiopulmonary exercise testing
* Weight > 190 kg (due to weight restrictions of equipment used to transfer patients in the event of medical emergencies)
* Cognitive impairment
* Patients unable to follow instructions in English

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with scheduled bariatric surgery at St George's Healthcare NHS Trust.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2014-06; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Cardiorespiratory function assessed by peak oxygen consumption (VO2peak) | One to two weeks before surgery and six months after surgery

SECONDARY OUTCOMES:
Lung function | One to two weeks before surgery and six months after surgery
  Lung function will be assessed by spirometry and body plethysmography
Heart function | One to two weeks before surgery and six months after surgery
  Echocardiography will be performed to assess heart function.
Inspiratory muscle strength | One to two weeks before surgery and six months after surgery
  Maximal inspiratory pressure and sniff nasal pressure will be recorded.
Peripheral muscle strength | One to two weeks before surgery and six months after surgery
  Maximum isometric strength of hand/ forearm, quadriceps and hip flexors muscles will be evaluated
Free living sedentary and physical activity times | One to two weeks before surgery and six months after surgery
  Daily physical activity habits will be assessed by an accelerometer and International Physical Activity Questionnaire: Long (IPAQ-Long). Participants will be required to wear the accelerometer for four consecutive days during the two study points.

CONTACTS AND LOCATIONS:
Overall Officials: Marcia S Volpe, Principal Investigator — Universidade Federal Triangulo Mineiro; Dimitra Nikoletou, Study Chair — Kingston University and St George's University of London; Marcus Reddy, Study Director — St George's Healthcare NHS Trust
Locations (1):
- St George's Healthcare NHS Trust, London, United Kingdom